CLINICAL TRIAL: NCT01688141
Title: A Primary-Secondary Care Partnership to Prevent Adverse Outcomes in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Shelton
Record Dates: First submitted 2009-11-20; First posted 2012-09-19 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease
Keywords: CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care
- Enhanced Management (Active Comparator): Practices randomised to the intervention group will be offered an enhanced level of CKD disease management led by clinical nurse specialists based on an intervention previously piloted in high risk patients. Here, high risk patients identified will be invited to a CKD clinic for tailored management of bp and proteinuria and referral as needed.
  Interventions: Other: Enhanced management

INTERVENTIONS:
Other: Enhanced management — Specialist nurses providing enhanced CKD management using NICE guidelines and enhanced access to secondary care.
  Other Names: CKD management
  Arms: Enhanced Management

SUMMARY:
Chronic kidney disease (CKD) is a major public health problem with a UK prevalence of 8-10%. The study hypothesis is to ascertain if intensive primary care led disease management programmes for CKD, supported by input from secondary care specialists will slow progression of CKD, improve blood pressure control and reduce cardiovascular events in patients on CKD registers.

The investigators have partnered with Nene commissioning, a practice based commissioning group representing approximately 80 GP practices in Northamptonshire, to run this study. This will be a cluster randomised trial of an intensive, secondary care supported, CKD management programme in primary care vs normal CKD care. Randomisation will be at the level of the individual general practice. All general practices associated with Nene commissioning will be invited to participate. Randomisation of practices will be performed by the University of Leicester Clinical Trials Unit and the study will adhere to guidelines for undertaking randomised cluster trials.

The aims of the study are:

1. To determine whether reinforcement of best practice in the management of key aspects of CKD care by clinical nurse specialists based in primary care, but with close links to colleagues from secondary care, improves clinical outcomes.
2. To foster excellence in CKD care
3. To improve coding of CKD and prevalence on chronic disease registers.
4. To increase interest in, and capacity for primary care research in Northamptonshire.
5. To implement and evaluate a new model of partnership working between primary and secondary care.

The primary outcome measures will be changes in estimated glomerular filtration rate (eGFR). Secondary outcome measures will be blood pressure control, proteinuria, incidence of cardiovascular events,other biochemical parameters, referrals to secondary care and hospitalisations and mortality.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* measurement of serum creatinine
* eGFR < 60 ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28304 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Brunskill, PhD, Principal Investigator — Consultant
Locations (3):
- United Kingdom (3):
  - Leicester General Hospital, Leicester, Leics
  - University Hospitals Leicester, Leicester, Leics
  - University Hospitals of Leicester, Leicester

REFERENCES:
- [Background] Major RW, Brown C, Shepherd D, Rogers S, Pickering W, Warwick GL, Barber S, Ashra NB, Morris T, Brunskill NJ. The Primary-Secondary Care Partnership to Improve Outcomes in Chronic Kidney Disease (PSP-CKD) Study: A Cluster Randomized Trial in Primary Care. J Am Soc Nephrol. 2019 Jul;30(7):1261-1270. doi: 10.1681/ASN.2018101042. Epub 2019 May 16. PMID 31097609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Enhanced Management
Started | 11706 | 11651
Completed | 11706 | 11651
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Enhanced Management | Total
Number analyzed (Participants) | 11706 | 11651 | 23357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 11706 | 11651 | 23357
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (11.3) | 75.1 (11.4) | 75.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7285 | 7234 | 14519
  Male | 4421 | 4417 | 8838
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11706 | 11651 | 23357

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean CKD Register Patient eGFRs Between Groups After 3.5 Years of Study
Time Frame: Baseline and 3.5 years
Measure: Mean (95% Confidence Interval); unit: mean average eGFR change/mL/min/1.73 m^2
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 11706 | 11651
mean average eGFR change/mL/min/1.73 m^2 | -2.00 [-3.95 to 0.92] | -2.29 [-3.89 to -0.69]

2. Secondary Outcome: Blood Pressure Control
Description: Observation of blood pressure control over the study period via blood pressure targets
Time Frame: Baseline and 3.5 years
Population: Denominator change due to loss to follow-up and death.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 11551 | 11473
Participants
  Baseline | 6834 | 7137
  3.5 Years: number analyzed (Participants) | 11129 | 10689
  3.5 Years | 7460 | 7295

3. Secondary Outcome: Proteinuria
Description: Proteinuria coding in practices
Time Frame: 3.5 years
Population: Loss to follow-up and death
Measure: Number; unit: participants
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 11689 | 11546
participants
  Baseline | 627 | 982
  3.5 Years: number analyzed (Participants) | 11228 | 10755
  3.5 Years | 1947 | 2110

4. Secondary Outcome: Incidence of Cardiovascular Events
Description: Observation of incidence of cardiovascular events over the study period
Time Frame: 3.5 years
Population: Data not available for analysis.
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Other Biochemical Parameters
Description: Nature and incidence over the study period
Time Frame: 3.5 years
Population: Data not available for analysis.
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Referrals to Secondary Care and Hospitalisations
Description: Data coillected from secondary care
Time Frame: 3.5 years
Population: Data not available for analysis.
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mortality
Description: data collected from secondary care
Time Frame: 3.5 years
Population: Data not available for analysis.
Arm/Group | Control | Enhanced Management
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Enhanced Management
Serious Adverse Events (participants affected / at risk) | 0/11706 | 0/11651
Other Adverse Events (participants affected / at risk) | 0/11706 | 0/11651

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No